CLINICAL TRIAL: NCT06518174
Title: A Novel Imaging Modality to Evaluate Radiation-Induced Uterine Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-5074.cc
Record Dates: First submitted 2024-07-08; First posted 2024-07-24 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Uterine Injury
Keywords: Uterine Injury; Radiation
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cases undergone PRT (Active Comparator): Patients (or their legal guardians) who opt for participating in this pilot study will be consented and enrolled in the study. Patients will then be scheduled for a single study visit at the University of Colorado Hospital (UCH) that includes:
  1. Pregnancy test
  2. Pelvic MRI without and with contrast (if patient consents to contrast)
  3. Transabdominal pelvic ultrasound using standard B-mode and Doppler US, SWE
  4. Optional transvaginal ultrasound using standard B-mode and Doppler US, SWE
  Interventions: Diagnostic Test: MRI, SWE, and US evaluation
- Controls (Sham Comparator): Controls (or their legal guardians) who opt for participating in this pilot study will be consented and enrolled in the study. Patients will then be scheduled for a single study visit at the University of Colorado Hospital (UCH) that includes:
  1. Pregnancy test
  2. Pelvic MRI without and with contrast (if patient consents to contrast)
  3. Transabdominal pelvic ultrasound using standard B-mode and Doppler US, SWE
  4. Optional transvaginal ultrasound using standard B-mode and Doppler US, SWE
  Interventions: Diagnostic Test: MRI, SWE, and US evaluation

INTERVENTIONS:
Diagnostic Test: MRI, SWE, and US evaluation — We will perform SWE and MRI sampling of the uterus from fundus to lower uterine segment with at least two points each from the upper, mid, and lower thirds of the uterus. SWE and MRI will be performed at time of study recruitment. US procedures will be transabdominal. When possible, we will also collect transvaginal US. MRI images will also be sampled from existing pretreatment studies performed as standard of care. All images will be evaluated for the presence and degree of fibrosis. We will compare SWE and MRI post-treatment. We will also compare pre-and post-treatment MRI.
  We will perform US and estimate uterine volumes and arterial resistance. Use descriptive statistics to compare values to age-matched controls

SUMMARY:
The goal of this pilot study is to assess the ability of a new imaging modality, shear-wave-elastography (SWE) and magnetic resonance imaging (MRI) to identify radiation-induced uterine injury (RIUI). The investigator will recruit female patients treated before 40 years with pelvic radiation (PRT) at least 12 months prior to study initiation.

DETAILED DESCRIPTION:
The investigator will recruit female patients treated before 40 years with pelvic radiation (PRT) at least 12 months prior to study initiation.12 months is selected to increase the occurrence of uterine fibrosis. The investigator will perform transabdominal standard B-mode and Doppler US, SWE and pelvic MRI and characterize uterine parameters. The B-mode and Doppler US will be referred to collectively as US. This will provide essential information to design an intervention trial of a novel therapeutic approach to the treatment of radiation-induced uterine damage. The overall objective of the study will be achieved through the following specific aims:

Aim 1: Assess the feasibility of SWE and pelvic MRI to identify and characterize uterine fibrosis. Hypothesis: A grid map sampling of the uterus will indicate feasibility of SWE and pelvic MRI to detect and characterize uterine fibrosis.

Approach: SWE and MRI will be performed at time of study recruitment. US procedures will be transabdominal. When possible, and with participant consent, transvaginal US will also be performed. MRI images will also be sampled from existing pretreatment studies performed as standard of care.

Perform SWE and MRI sampling of the uterus from fundus to lower uterine segment at two locations each from the upper, mid, and lower thirds of the uterus (six grid sample locations).

Obtain five measurements at each location to evaluate for the presence and degree of fibrosis:

1. Assess the relationship between SWE measurements in kiloPascals (kPa) and each MRI parameter among cases at the post-treatment timepoint.
2. Assess the relationship between SWE measurements and each MRI parameter in kPa among controls at one random timepoint.
3. Evaluate differences in kPa between cases and controls according to SWE at the post-treatment timepoint. The imaging study will be considered feasible if at least 85% (e.g., ≥15/17) of all enrolled cases achieve the diagnosability criteria by SWE, defined as having the interquartile range to median ratio (IQR/M) of the measurements (kPa) <=30% at any of the six locations.

Aim 2: Characterize uterine parameters after PRT. Hypothesis: Patients treated with PRT for colorectal/anal cancer will have decreased uterine volume and increased arterial resistive indices (blood flow) on US.

Approach:

2a. Perform US and estimate uterine volumes and arterial resistance. Use descriptive statistics to compare values to controls in the same age group.

2b. Perform MRI and describe changes in each parameter among cases between the pre- and post-treatment timepoints. Assess changes in: size of the uterus from baseline, junctional zone anatomy, endometrial thickness, cervical length, myometrial thickness, T2 signal of the myometrium (normalized for skeletal muscle signal acting as an internal control), and enhancement features.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Less than 40 years old "at the time of pelvic radiation"
3. ≥ 18 and < 45 years of age "at time of enrollment"
4. Treated with PRT at UCH
5. Pelvic MRI taken before the pelvic radiation

Exclusion Criteria:

1. Patients who underwent hysterectomy for treatment of a primary gynecologic malignancy
2. Patients that are currently pregnant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 22 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
SWE feasibility | Up to six months
  SWE will be considered feasible if at least 85% (e.g., ≥15/17) of all patients achieve the diagnosability criteria, defined as having at least 1 of 6 locations with IQR/M ≤ 30%. The IQR/M and the number of patients who achieved diagnosability will be descriptively characterized.
Compare the degree of fibrosis according to SWE and MRI parameters across treatment groups | Up to six months
  Since fibrosis thresholds have not been thoroughly established for SWE tissue stiffness nor MRI parameters, continuous SWE tissue stiffness (kPA) will be compared separately to each MRI parameter: uterus size, junctional anatomy, endometrial thickness, cervical length, myometrial thickness, T2 signal, and enhanced features.
Evaluate the correlation between MRI images collected at pretreatment and after recruitment, using repeated measures correlation. | Up to six months
  Descriptive statistics and previously described figures will be similarly used to characterize the change in each MRI parameter between the pre-treatment and post-treatment timepoints. Additionally, linear mixed effects regression models will be performed separately with each MRI parameter. The predictors will include pre- and post- treatment time points and treatment group. If appropriate, radiation dose will be included in the model as well, where the radiation dose will be assigned as 0 for the control patients. Contrast statements will be used to assess the change in each outcome comparing treatment groups and the radiation doses effect.

SECONDARY OUTCOMES:
Characterize uterine parameters after PRT | Up to six months
  On-study uterine volume and arterial resistance will then be assessed with SWE. Previously described descriptive statistics and plots will be used to depict differences in each measurement across cases and controls. Sample size permitting, t-tests will be considered to secondarily quantify the differences across groups. Transabdominal and transvaginal SWE measurements will also be compared as an exploratory endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Milgrom, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States